CLINICAL TRIAL: NCT04616846
Title: Thromboembolic Risk Screening in Patients With Cancer and COVID-19
Acronym: NEOTHROCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 2020/20
Record Dates: First submitted 2020-11-02; First posted 2020-11-05 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Neoplasms Malignant; Covid19; Thromboembolism
Keywords: cancer; Covid19; Thromboembolism
MeSH Terms: conditions — Neoplasms; COVID-19; Thromboembolism

STUDY DESIGN:
Intervention Model Description: Retrospective and prospective (ambispective), multicentric study to evaluate the occurrence of venous thromboembolism during COVID-19 infection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control cohort (No Intervention)
- Infected cohort (Experimental)
  Interventions: Diagnostic Test: Peripheral venous ultrasound

INTERVENTIONS:
Diagnostic Test: Peripheral venous ultrasound — Screening for VTE from D7 to 42
  Arms: Infected cohort

SUMMARY:
Study Rational

Since December 2019, outbreak of COVID-19 caused by a novel virus SARS-Cov-2 has spread rapidly around the world and became a pandemic issue. First data report high mortality in severe patients with 30% death rate at 28 days. Exact proportions of the reasons of death are unclear: severe respiratory distress syndrome is mainly reported which can be related to massive cell destruction by the virus, bacterial surinfection, cardiomyopathy or pulmonary embolism. The exact proportion of all these causes is unknown and venous thromboembolism could be a major cause because of the massive inflammation reported during COVID-19.

High levels of D-dimers and fibrin degradation products are associated with increased risk of mortality and some authors suggest a possible occurrence of venous thromboembolism (VTE) during COVID-19.

Indeed, COVID-19 infected patients are likely at increased risk of VTE. In a multicenter retrospective cohort study from China, elevated D-dimers levels (>1g/L) were strongly associated with in-hospital death, even after multivariable adjustment.

Also, interestingly,the prophylactic administration of anticoagulant treatment was associated with decreased mortality in a cohort of 449 patients, with a positive effect in patients with coagulopathy (sepsis-induced coagulopathy score ≥ 4) reducing the 28 days mortality rate (32.8% versus 52.4%, p=0.01).

However the presence/prevalence of VTE disease is unknown in COVID-19 cancer patients with either mild or severe disease. Cancer patients are at a higher risk of VTE than general population (x6 times) and could be consequently at a further higher of VTE during COVID-19, in comparison with non-cancer patients.

The exact rate of VTE and pulmonary embolism during COVID-19 was never evaluated, especially in cancer patients, and is of importance in order to understand if this disease needs appropriate prophylaxis against VTE.

The largest series of cancer patients so far included 28 COVID-19 infected cancer patients: the rate of mortality was 28.6%. 78.6% of them needed oxygen therapy, 35.7% of them mechanical ventilation. Pulmonary embolism was suspected in some patients but not investigated due to the severity of the disease and renal insufficiency, reflecting the lack of data in this situation.

The aim of the present study is to analyze the rate of symptomatic/occult VTE in a cohort of patients with cancer.

Expected benefits Anticipated benefits of the research are the detection of VTE in order to treat it for the included patient.

For all COVID-19 positive cancer patients it will enable to provide some guidelines and determine which patient are at risk for VTE and which will need ultrasound to detect occult VTE.

Foreseeable risks Foreseeable risks for patients are non-significant because the additional procedures needed are ultrasound exam, and blood sample test.

Methodology

Retrospective and prospective (ambispective), multicentric study to evaluate the occurrence of venous thromboembolism during COVID-19 infection.

Indeed, because the outbreak can end within the next 3-6 months, Investigators may not be able to answer the question if Investigators only focus on patients investigated prospectively. Investigators then decided to include patients from medical team who are already systemically screening patients with COVID-19 disease for VTE.

Trial objectives

Main objective To evaluate the rate of venous thromboembolism at 23 days during COVID-19 infection in cancer patients.

DETAILED DESCRIPTION:
Study Rational

Since December 2019, outbreak of COVID-19 caused by a novel virus SARS-Cov-2 has spread rapidly around the world and became a pandemic issue. First data report high mortality in severe patients with 30% death rate at 28 days. Exact proportions of the reasons of death are unclear: severe respiratory distress syndrome is mainly reported which can be related to massive cell destruction by the virus, bacterial surinfection, cardiomyopathy or pulmonary embolism. The exact proportion of all these causes is unknown and venous thromboembolism could be a major cause because of the massive inflammation reported during COVID-19.

High levels of D-dimers and fibrin degradation products are associated with increased risk of mortality and some authors suggest a possible occurrence of venous thromboembolism (VTE) during COVID-19.

Indeed, COVID-19 infected patients are likely at increased risk of VTE. In a multicenter retrospective cohort study from China, elevated D-dimers levels (>1g/L) were strongly associated with in-hospital death, even after multivariable adjustment.

Also, interestingly, the prophylactic administration of anticoagulant treatment was associated with decreased mortality in a cohort of 449 patients, with a positive effect in patients with coagulopathy (sepsis-induced coagulopathy score ≥ 4) reducing the 28 days mortality rate (32.8% versus 52.4%, p=0.01).

However the presence/prevalence of VTE disease is unknown in COVID-19 cancer patients with either mild or severe disease. Cancer patients are at a higher risk of VTE than general population (x6 times) and could be consequently at a further higher of VTE during COVID-19, in comparison with non-cancer patients.

The exact rate of VTE and pulmonary embolism during COVID-19 was never evaluated, especially in cancer patients, and is of importance in order to understand if this disease needs appropriate prophylaxis against VTE.

The largest series of cancer patients so far included 28 COVID-19 infected cancer patients: the rate of mortality was 28.6%. 78.6% of them needed oxygen therapy, 35.7% of them mechanical ventilation. Pulmonary embolism was suspected in some patients but not investigated due to the severity of the disease and renal insufficiency, reflecting the lack of data in this situation.

The aim of the present study is to analyze the rate of symptomatic/occult VTE in a cohort of patients with cancer.

Expected benefits Anticipated benefits of the research are the detection of VTE in order to treat it for the included patient.

For all COVID-19 positive cancer patients it will enable to provide some guidelines and determine which patient are at risk for VTE and which will need ultrasound to detect occult VTE.

Foreseeable risks Foreseeable risks for patients are non-significant because the additional procedures needed are ultrasound exam, and blood sample test.

Methodology

Retrospective and prospective (ambispective), multicentric study to evaluate the occurrence of venous thromboembolism during COVID-19 infection.

Indeed, because the outbreak can end within the next 3-6 months, Investigators may not be able to answer the question if Investigators only focus on patients investigated prospectively. Investigators then decided to include patients from medical team who are already systemically screening patients with COVID-19 disease for VTE.

Trial objectives

Main objective To evaluate the rate of venous thromboembolism at 23 days during COVID-19 infection in cancer patients.

Secondary objectives

The secondary objectives are:

1. To determine the 23-days rate of hospitalization due to venous thromboembolism;
2. To determine the 23-days Overall Survival (OS);
3. To determine the 23-days Specific Survival (SS, death due to venous thromboembolism);
4. To evaluate the global safety of antineoplastic treatment;
5. To determine the predictive factors of venous thromboembolism;
6. To compare the rate of symptomatic venous thromboembolism between the COVID-19 negative and COVID-19 positive patients.

Ancillary study Collection of blood sample in order to detect thrombophilia in case of venous thromboembolism.

Description of specifics procedure

For the prospective cohort:

Day 1 = Day when COVID-19 test is performed.

* Blood sample (Day 1 for every patient tested for COVID19 infection) three 1.8ml citrate tubes, three 3ml Heparin and two 4 ml EDTA tubes:
* Count of Hb, platelet, leukocytes, neutrophils, lymphocytes,
* LDH, CRP, Procalcitonin, D-dimers, ferritin, fibrin degradation product, sodium, potassium, ASAT, ALAT, GGT, PAL, TP, TCA,
* Bilirubin, calcium, protein, albumin, fibrinogen, troponin, BNP.
* 2 Peripheral venous Ultrasound (if positivity for COVID19 and if positive D-dimers, at day 1-10 after diagnosis and day 20-23):
* analysis of femoral, popliteal, tibial and peroneal venous,
* analysis of venous where there is material/central catheters,
* analysis of any venous where there is symptom of VTE.
* ECG (the day of peripheral venous ultrasound)
* Computed-tomography scan with iodin contrast injection: if suspicion of pulmonary embolism
* Transthoracic ultrasound (the day of peripheral venous ultrasound): if pulmonary emboly signs and no availability or possibility to do computed-tomography scan: clinical emboly sign are dyspnea, hemoptysis, chest pain, tachycardia, palpitations, ECG signs.
* Ancillary study = thrombophilia analysis if occurrence of VTE, five 10ml citrate tubes and two 10 ml EDTA tubes : anti-thrombin 3, protein S deficit, protein C deficit, homocystein, circulating anticoagulant, Antibody against beta 2 gp1, Antibody against cardiolopin, Activated protein C resistance, mutation of Factor V and II of Leiden. The thrombophilia analysis, as part of the routine practice, will be also performed in the retrospective cohort and if occurrence of VTE.
* For patient negative for COVID-19 infection, a second test will be performed between Day20-Day23 to confirm the negativity of COVID-19 exposure.

Of note: dedicated ultrasound device will be used only for COVID-19 infected patients.

Statistical analysis plan

All statistical analyses will be performed at alpha risk=5% in bilateral hypothesis by the statistician of the Center Antoine Lacassagne using R.3.6 and SAS 9.4 software for windows.

The cumulative rate of VTE is about 2-4% over a period of 70 days in patients treated for cancer and at the start of chemotherapy.

Major well known risk factors for VTE are: certain type of cancer (stomach, pancreas, lung, lymphoma, gynecologic, genitourinary without prostate), body mass index ≥ 35, platelets count ≥ 350 000/mm3, Hemoglobin level < 10 gr/dL (or use of red cell growth factors), leucocyte cell count > 11 000/mm3. 27% of patients present with low risk Khorana score (score 0) that is 0.8% occurrence of VTE, 60.2% with intermediate risk (Khorana score of 1-2) that is 1.8% occurrence of VTE and 12.8% high risk (Khorana score ≥ 3) that is 7.1% risk of VTE. Of note the rate of occult VTE in patients with high risk is about 9% in a cohort of 35 patients.

The aim of the study is to describe the proportion of VTE in patients with cancer presenting a COVID-19 infection.

We estimate that forty patients are needed to have an appropriate overview of the incidence in COVID-19 patients. In order to compare with a similar non-infected cohort Investigators will also include patients with cancer tested negative for COVID-19 during the same period (as soon as possible, a serology will be used thereafter to confirm it). All patients with cancer tested negative for COVID-19 will be included. Investigators estimate that 80 patients are needed to have an appropriate overview of the rate of VTE in the control cohort. This negative cohort will be further tested with serology as soon as available, to check if they were tested as false negative.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 testing ;
* Age ≥ 18 years old ;
* Patient treated for histologically proven cancer (under treatment or last anti-neoplastic treatment < 3 months at the time of COVID-19 testing);
* For the infected cohort: patient being screened for VTE at least one time 7 weeks after the COVID-19 diagnosistwo time point (day 1-10 after COVID-19 testing, and day 20-25 after COVID-19 testing) for retrospective cohort only;
* Complete blood count available at time of COVID-19 testing (+/-14 days) to be able to calculate the Khorana score;
* Patient informed and not opposed to the data processing;
* Patient affiliated with a health insurance system.

Exclusion Criteria:

* Patient not able to give free consent;
* Patient not able to understand the protocol;
* For the infected patients: VTE screening not performed (for retrospective cohort only);
* No available complete blood count at time of COVID-19 testing; Medical file and clinical follow-up not available during the study period (76 weeks after the COVID-19 test);
* Patients under 18 years;
* Vulnerable persons as defined by article L1121-5-8:

  1. Pregnant women, women in labour or breast-feeding mothers, persons deprived of their freedom by judicial or administrative decision, persons hospitalized without their consent by virtue of articles L. 3212-1 and L. 3213-1 and who are not subject to the provisions of article L. 1121-8
  2. Persons admitted to a social or health facility for reasons other than research
  3. Adults subject to a legal protection order or unable to give their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Rate of venous thromboembolism | From Day 9 to Day 42
  Deep venous thrombosis and/or pulmonary embolism.

SECONDARY OUTCOMES:
Hospitalization due to venous thromboembolism | Day 23
  Rate of hospitalization
Overall Survival | Day 23
  Time between the date of inclusion and the date of death for any reason.
Specific survival | Day 23
  Time between the date of inclusion and the date of death for venous thromboembolism.
Safety profile using the common toxicity criteria from the NCI CTCAE V5.0 | Day 1 to Day 23
  Common toxicity criteria from the NCI CTCAE V5.0
Predictive factors for venous thromboembolism | Day 1 to Day 23
  Khorana score (low risk (score=0), medium risk (score=1 ou 2) and high risk (score ≥ 3)
Predictive factors for venous thromboembolism | Day 1 to Day 23
  Caprini score (very low risk (score=0), low risk (score=1 or 2), medium risk (score=3 or 4)and high risk (score ≥ 5)
rate of symptomatic venous thromboembolism between the COVID-19 negative and COVID-19 positive patients | Day 1 to Day 23
  Common toxicity criteria from the NCI CTCAE V5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme DOYEN, MD-PHD, Principal Investigator — Centre Antoine Lacassagne
Locations (6):
- France (5):
  - Clinique Saint-Jean, Cagnes-sur-Mer, Alpes-Maritimes
  - Centre Azuréen de Cancérologie, Mougins, Alpes-Maritimes
  - CHU Nice, Nice, Alpes-Maritimes
  - Clinique Saint-Georges, Nice, Alpes-Maritimes
  - Centre Antoine Lacassagne, Nice, Alpes-Maritimes
- CHPG, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No